CLINICAL TRIAL: NCT00514007
Title: A Phase I Dose Escalation Study of Continuous Oral OSI-906 Dosing in Patients With Advanced Solid Tumors
Brief Title: Study of Continuous OSI-906 Dosing
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSI-906-101; 2006-005937-39 (EudraCT Number)
Record Dates: First submitted 2007-08-07; First posted 2007-08-09 (Estimated); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Advanced Solid Tumors
Keywords: Advanced Cancer; Colorectal cancer; Ovarian cancer; Renal cancer; Metastatic cancer; Breast cancer; Non-small cell lung cancer
MeSH Terms: conditions — Colorectal Neoplasms; Ovarian Neoplasms; Kidney Neoplasms; Neoplasm Metastasis; Breast Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — 3-(8-amino-1-(2-phenylquinolin-7-yl)imidazo(1,5-a)pyrazin-3-yl)-1-methylcyclobutanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- OSI-906 QD (Experimental): Once per day
  Interventions: Drug: OSI-906
- OSI-906 BID (Experimental): Twice per day
  Interventions: Drug: OSI-906

INTERVENTIONS:
Drug: OSI-906 — OSI-906 administered orally

SUMMARY:
Multicenter, open-label, phase 1, cohort dose escalation study to determine the Maximum Tolerated Dose (MTD) on both Once Daily (QD) and Twice Daily (BID) schedules.

DETAILED DESCRIPTION:
Multicenter, open-label, phase 1, cohort dose escalation.

The study will open with the QD schedule, with initiation of the BID schedule occurring after observation of clinically significant related toxicity ≥ grade 2 in the QD schedule.

Dosing will be initiated on Day 1 with daily dosing (either QD or BID) continuing for 21 days.

Once the recommended phase 2 dose has been determined for the BID schedule, 2 expansion cohorts will be opened: 1) Biomarker Expansion Cohort in patients with locally advanced or metastatic colorectal cancer and 2) Diabetic Expansion Cohort in patients with advanced solid tumors who have active Type 2 diabetes mellitus not requiring insulin or insulinotropic therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically documented malignancy that is now advanced and/or metastatic and refractory to established forms of therapy or for which no effective therapy exists. Patients in the Biomarker Expansion Cohort must have histologically documented colorectal cancer that is locally advanced or metastatic and refractory to established forms of therapy. These patients must have archival tissue available and a lesion accessible for biopsy
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0-2, life expectancy ≥ 12 weeks
* Prior chemotherapy is permitted provided that a minimum of 3 weeks has elapsed. Prior tyrosine kinase inhibitor therapy is permitted. Patients must have recovered from any treatment-related toxicities (with some exceptions) prior to registration
* Prior hormonal therapy is permitted provided it is discontinued prior to registration (with the exception of prostate cancer patients who have been on hormone therapy for at least 3 months)
* Prior radiation therapy is permitted provided that patients have recovered from the toxic effects. A minimum of 21 days must have elapsed unless the radiotherapy was palliative and nonmyelosuppressive
* Prior surgery is permitted provided that wound healing has occurred prior to registration
* Fasting glucose ≤ 125 mg/dL (7 mmol/L) at baseline (all patients except those in the Diabetic Expansion Cohort). Patients in the Diabetic Expansion Cohort must have a fasting glucose of ≤ 150 mg/dL (8.3 mmol/L) at baseline. If patients in the Diabetic Expansion Cohort are being treated with non-insulinotropic oral antihyperglycemic therapy, doses must be stable for ≥ 4 weeks prior to registration
* Potassium, calcium, and magnesium must be within normal limits (WNL). Electrolyte abnormalities will be permitted if they are not clinically significant and if treatment for the abnormality is initiated prior to Day 1
* Neutrophil ≥ 1.5 x 10^9/L, Platelet (PLT) ≥ 100 x 10^9/L; bilirubin ≤ 1.5 x upper limit of normal (ULN), AST and ALT ≤ 2.5 x ULN or ≤ 5 x UNL if patient has documented liver metastases; creatinine ≤ 1.5 x ULN
* Accessible for repeat dosing and follow-up, including pharmacokinetic sampling
* Patients must practice effective contraceptive measures throughout the study
* Provide written informed consent

Exclusion Criteria:

* History of any kind of stroke
* History of any psychiatric condition that might impair the patient's ability to provide informed consent or participate
* History of allergic reaction attributed to a similar compound as study drug.
* Any type of active seizure disorder
* Previously diagnosed brain metastases
* Concurrent anticancer therapy
* Active or uncontrolled infections of serious illnesses or medical conditions that could interfere with participation
* Pregnant or breast-feeding females
* Documented history of diabetes mellitus (all patients except those in the Diabetic Expansion Cohort). Patients in the Diabetic Expansion Cohort may not have Type 1 diabetes mellitus or Type 2 diabetes mellitus currently requiring insulinotropic or insulin therapy
* Use of drugs with a risk of causing QT interval prolongation within 14 days prior to Day 1 and while on study
* Use of glucocorticoids within 14 days prior to Day 1 and while on study
* History of significant cardiac disease unless well controlled (includes 2nd/3rd degree heart block, ischemic heart disease, QTc > 450 msec, poorly controlled hypertension, or congestive heart failure of New York Heart Association (NYHA) Class II or worse)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2007-06-18 (Actual); Primary Completion 2012-03-19 (Actual); Study Completion 2012-03-19 (Actual)

PRIMARY OUTCOMES:
Determine the maximum tolerated dose (MTD) for both the once daily (QD) and twice daily (BID) dosing schedules and establish a recommended phase 2 dose of oral OSI-906 | 21 days

SECONDARY OUTCOMES:
Safety profile; Pharmacokinetic (PK) profile; Pharmacodynamic relationships and preliminary antitumor activity | 2.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Global Development
Locations (2):
- Vanderbilt Universtiy Medical Center, Nashville, Tennessee, United States
- The Beatson West of Scotland Cancer Centre, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- See also: Link to results on the Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=267